CLINICAL TRIAL: NCT02650167
Title: Impact of Oropharyngeal Administration of Colostrum in the First 48 Hours of Life Term Premature Newborn ≤ 32 Weeks of Amenorrhea
Acronym: COLOSTRUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15-AOI-02
Record Dates: First submitted 2016-01-06; First posted 2016-01-08 (Estimated); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Infant, Premature
MeSH Terms: conditions — Premature Birth | interventions — Food, Formulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colostrum (Experimental)
  Interventions: Biological: Colostrum feeding
- Witness (Experimental)
  Interventions: Biological: formula for preterm infants

INTERVENTIONS:
Biological: Colostrum feeding
  Arms: Colostrum
Biological: formula for preterm infants
  Arms: Witness

SUMMARY:
Colostrum is the first milk secreted by the mother when the tight junctions of mammary epithelium open, allowing the cellular transport of a multitude of components and immunological protective derivatives of the maternal circulation to the milk, and especially immunoglobulins A type. Colostrum is not given to preterm neonates. The assumption behind this work is that the oro pharyngeal administration of colostrum early in preterm infants could help deliver an oral immunotherapy even before the installation of enteral nutrition, through interactions with lymphoid tissues of the oropharynx and the gastrointestinal tract. This practice would improve the digestive tolerance and the establishment of enteral feeding, the decrease in mucosal inflammatory phenomena, but also to provide any protection against subsequent infections. Finally, there could be an improvement in the secondary immune tolerance with a decrease in the occurrence of allergic phenomena.

ELIGIBILITY:
Inclusion Criteria:

* New premature infant with a term weight ≤ 32 weeks amenorrhea at Nice University Hospital
* Mother seronegative for HIV

Exclusion Criteria:

* Neonates with congenital pathologies immediate prenatal or neonatal diagnosis will not be included.
* Therapy of the mother incompatible with breastfeeding during pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-04-27 (Actual); Primary Completion 2018-05-05 (Actual); Study Completion 2020-09-24 (Actual)

PRIMARY OUTCOMES:
Measuring caloric intake (number of days required for the calorie intake) | 2 days
  number of days required for the calorie intake to 130 kcal / kg / day can be delivered exclusively enterally

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie DE SMET, Dr, Study Director — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France